CLINICAL TRIAL: NCT06254963
Title: The Effect of 6 Weeks Supplemental Jump Training on Sand Versus Hard Surfaces on Landing Knee Valgus and Jump Performance in Adolescent Female Football Players
Brief Title: The Effect of 6 Weeks Jump Training on Sand Versus Hard Surfaces on Jump Landing and Performance in Young Females
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Teesside University (Other)
Collaborators: University of Sunderland (Other)
Responsible Party: Principal Investigator, Mark Richardson, Senior Lecturer, Allied Health Professions Department, Teesside University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Jan24 18946
Record Dates: First submitted 2024-02-02; First posted 2024-02-12 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Frontal Plane Projection Angle; Maximal Countermovement Jump; Repeated 10/5
Keywords: sand; jump training; knee valgus; jump height

STUDY DESIGN:
Intervention Model Description: Participants will be randomised into one of 2 groups, either supplemental sand jump training or land jump training.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sand jump training (Experimental): Participants will conduct 6 weeks (twice weekly) supplemental jump training on a sand surface (within their warm ups) in addition to their regular training.
  Interventions: Other: sand jump training
- Land jump training (Active Comparator): Participants will conduct 6 weeks (twice weekly) supplemental jump training on a land surface (within their warm ups) in addition to their regular training.
  Interventions: Other: land jump training

INTERVENTIONS:
Other: sand jump training — A series of progressive jumping activities on sand increasing in difficulty over the 6 week period
  Arms: Sand jump training
Other: land jump training — A series of progressive jumping activities on land increasing in difficulty over the 6 week period
  Arms: Land jump training

SUMMARY:
The aim of this study is to investigate the effect of a supplemental jump training program (added to a warm up) conducted on either sand or hard surfaces on the landing and jumping ability of young female football players. The jump training program (intervention) will be carried out twice weekly for a period of 6 weeks. Participants will be randomised (computer package will decide) into one of 2 groups (either sand training or land training). The landing ability and jumping performance of all participants will be measured both before and after the 6 week jump training intervention. It is hypothesised that supplemental training on both sand and hard surfaces will improve landing ability and jumping performance. It is also hypothesised that sand will be equally as effective as a hard surface for improving jump landing ability but may be less effective than a hard surface for improving jumping performance.

DETAILED DESCRIPTION:
Participants will be under 16 females currently training and playing for the football Emerging Talent Centre (ETC) at Teesside University.

The testing will take place at Teesside University. Participants will attend on 2 occasions (Pre and post intervention). During the first session participants age, height, and weight, will be collected. Participants will then perform a warmup consisting of fundamental movements like squatting, lunging, running, skipping and jumping.

Participants will then be asked to perform 5 practice trials of a single leg step landing task from a 30cm box. This will be demonstrated to them initially and then the practice trials will allow participants a chance to orient themselves to the task before data collection. For the step down task participants will be instructed to stand on the box and then step off the box and land and hold the position on their dominant leg (which is decided by the leg they prefer to kick a ball with).

Throughout testing participants will be required to wear reflective markers (14mm) over dark coloured shorts and top. The markers will be attached with double sided adhesive tape to the participants lower extremities over the following landmarks: anterior superior iliac spine (left and right), mid tibiofemoral joint (left and right) and mid talocrural joint (left and right). The same individual (MR) will place the markers on all participants. Midpoint will be determined using a standard tape measure. These markers will be used to calculate a knee angle on landing (specific outcome measure detailed elsewhere), measured using a high speed digital video camera (Quintic GigE 1mp; Quintic Consultancy Ltd, West Midlands, United Kingdom) recording at 200 frames per second, positioned 2 m anterior to the subjects' landing target at the height of the participant's knee and aligned perpendicular to the frontal plane. Images captured will be imported into a digitizing software program (Quintic 29; Quintic Consultancy Ltd) ready for analysis. The average landing value from 5 trials during the task will be used for analysis.

Following completion of the step-down task participants will then be asked to complete two performance tests (with a standardised 3 minute rest period between them). As within the step landing task they will be given practice trials to help familiarise themselves with the tests prior to data collection. The first test with be a countermovement jump (CMJ), where participants will stand on a force platform (built into the laboratory floor). Each foot will be on an individual force plate. Participants will then be asked to squat down, keeping their hands on their hips and subsequently jump as high as they can. Whilst in flight they must keep their hands on their hips and keep their leg straight. Participants will be instructed to land in the same position they took off from (i.e. not forward or backwards). Tape will be stuck on the floor as a marker to help guide the participants towards achieving this. The participant will perform 3 efforts with the average height being used for analysis. The second test is the 10/5 repeated jump test to evaluate the participants reactive strength index. The test requires the participant to execute 10 maximal rebound jumps (attempting to minimise ground contact time between jumps). Of the 10 jumps, the 5 that display the greatest jump height are used for analysis. The 10/5 test will be measured using the same in-ground force plate noted for the CMJ test. As with the CMJ test participants will be instructed to keep their hands on their hips throughout the jump phase and each of the 10 repeated jumps. One trial of the test is all that is required for data analysis purposes.

The testing protocol will be performed by all participants (pre and post an intervention time period of 6 weeks). There will be 2 groups (see below). Participants will be randomised into one of two groups. Both groups will perform a jump training protocol (on either a firm or sand surface) which involves a series of exercises that will be added to their usual warm up routine pre training. All participants will continue to train and play as normal during the intervention time period. They will then be invited back in at the end of the 6 week period for a second and final testing session.

The jump training protocol will involve a series of jumping tasks, which will be increased in difficulty level over the 6 week intervention period. The supplemental jump training protocol should take approximately 5-10 minutes to complete and will be incorporated into the participants warm up routine for their regularly training sessions x 2 weekly. Participants will continue with the rest of their football training as normal across the 6-week period.

ELIGIBILITY:
Inclusion Criteria:

* female under the age of 16 and have been deemed medically fit to train and play football by the Emerging Talent Centre
* parental consent and child assent gained
* no history of anterior cruciate ligament (ACL) injury or previous lower limb fracture or surgery
* no lower limb injury in the last 3 months.
* no allergy to hypoallergenic adhesive tape.

Exclusion Criteria:

* male
* 16 or over
* no parental consent and/or no child assent given
* not deemed medically fit to train and play football by the Emerging Talent Centre
* history of anterior cruciate ligament (ACL) injury or previous lower limb fracture or surgery
* lower limb injury in the last 3 months
* allergy to hypoallergenic adhesive tape

Ages: 10 Years to 15 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2024-02-14 (Actual); Primary Completion 2024-04-19 (Actual); Study Completion 2024-04-19 (Actual)

PRIMARY OUTCOMES:
Frontal Plane Projection Angle | 1 week pre intervention and 1 week post intervention
  The angle of knee valgus or varus upon landing
Maximal Countermovement Jump | 1 week pre intervention and 1 week post intervention
  Measure of jump height
10/5 Repeated Jump Test | 1 week pre intervention and 1 week post intervention
  Measures Reactive Strength Index

CONTACTS AND LOCATIONS:
Overall Officials: Mark C Richardson, MSc, Principal Investigator — Teesside University
Locations (1):
- Teesside University, Middlesbrough, Tees Valley, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
There is no specific plan to make IPD available at present but relevant data can be made available to other researchers following publication at reasonable request